CLINICAL TRIAL: NCT06803433
Title: Comparison Between Effectiveness of Different Esthetic Orthodontic Appliances in Management of Lower Anterior Teeth Relapse: a Randomized Clinical Trial
Brief Title: Comparison Between Effectiveness of Different Esthetic Orthodontic Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Assem Gamaleldin Esmat Mohamed Gamil, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-3-2
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Relapse of the Lower Anterior Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aligners (Experimental): The upper and lower arches will be intra orally scanned followed by fabrication of in office aligners for the lower arch using 3shape software.
  Interventions: Device: Aligners
- Lingual braces (Experimental): 2D lingual braces will be indirectly bonded to the lower anterior teeth from canine to canine.
  Interventions: Device: Lingual braces
- Active fixed lingual wire (Active Comparator): A customized 14 nickel-titanium archwire was placed on the lingual surfaces of the lower anterior teeth and secured through ligature wires passing through the contact points.
  Interventions: Device: Active fixed lingual wire

INTERVENTIONS:
Device: Aligners — Lower arch in office aligners.
  Arms: Aligners
Device: Lingual braces — Lingual braces bonded to the lower anterior teeth
  Arms: Lingual braces
Device: Active fixed lingual wire — A customized 14 Niti lingual wire customized to the lingual surface of the lower anterior teeth and secured with ligature wires.
  Arms: Active fixed lingual wire

SUMMARY:
The purpose of this study is to compare the effectiveness of active fixed lingual wire, removable aligners, and lingual braces in managing crowding of the lower anterior teeth resulting from relapse. The study intends to evaluate these interventions concerning the degree of alignment achieved in the lower anterior teeth, treatment duration, patient discomfort, patient acceptance, gingival inflammation and the cost effectiveness.

DETAILED DESCRIPTION:
1. Background Orthodontic relapse can be defined as the tendency for teeth to return to their pre- treatment position and this particularly occurs in the lower anterior teeth. Retention, to maintain teeth in their corrected position, has become one of the most important phases of orthodontic treatment, however, studies have revealed that the long-term alignment of the lower front teeth following orthodontic treatment was unsatisfactory. Post-treatment alignment (assessed by Little's irregularity index) may be maintained in only 30% to 50% of orthodontic patients over 10 years.

   Certain critical factors may contribute to the relapse of the lower front teeth. These include reorganization of the periodontal tissue, decrease of the crestal alveolar bone level, over- expansion of the arch dimension, occlusal changes due to mandibular growth, eruption of the third mandibular molars, type of malocclusion being treated and adverse effects of tooth movement during treatment.

   While labial braces may be the most effective method to correct relapse of lower front teeth, their use may be undesirable as patients may be reluctant to go through the experience of fixed brackets again.

   Active fixed lingual wire, removable aligners and fixed lingual braces are considered esthetic options to manage such condition. Aligners may address the demand for an esthetic alternative but could prove to be an expensive option and patient cooperation is mandatory. Fixed lingual braces may be more effective in correcting the relapse but their use may be undesirable due to speech problems, and tongue irritability.

   A recent cochrane systematic review assessing the the effects of interventions used to manage relapse of the lower front teeth stated that there is a need for rigorously conducted, and reported, RCTs to be undertaken to assess the effects of different approaches to orthodontic re- treatment following relapse of lower front teeth alignment.
2. Research Hypothesis:

   The null hypothesis for the study was that removable aligners, lingual braces and active fixed lingual wire have the same efficiency in managing relapse of lower anterior teeth in adult female patients.
3. Objectives:

Primary Objective:

The primary objective of this study is to evaluate the resolution of lower anterior teeth crowding by measuring the mean change in Little's Irregularity Index, which is defined as the sum of the linear distances between the anatomical contact points of the mandibular incisors.

Secondary Objectives:

To determine if aligners, lingual braces, and active fixed lingual wire will be able to:

* Resolve lower anterior teeth crowding by achieving a clinically acceptable Little's Irregularity Index of less than 1 mm within the treatment duration.
* Provide a well-accepted treatment experience based on patient-reported outcomes related to oral hygiene, pain, and discomfort.
* Minimize patient discomfort by assessing pain levels at multiple time points using a visual analog scale from 0 to 10.
* Maintain gingival health by evaluating gingival inflammation through the Gingival Index at different stages of treatment.
* Establish a cost-effective treatment modality by analyzing the cost-effectiveness of each intervention.

  4- Study design

According to the norms of the CONSORT STATEMENT, this study will be clinical with intervention, in which the allocation of the subjects will be randomized. This study will be parallel with blinding for the outcome assessors. The primary purpose of this study will be treatment.

5- Participants - Settings and locations where the data are collected

The treatment will be performed in the outpatient clinics of Department of Orthodontics of Cairo University. Data will be collected from June 2021 through February 2022.

6. Interventions Three groups will receive treatment. Group 1 will be treated with the Aligners for 6 months or until reaching a clinically acceptable little irregularity index of less than 1 mm. Group 2 will be treated with Lingual braces for 6 months or until reaching a clinically acceptable little irregularity index of less than 1 mm. Group 3 will be treated with the active fixed lingual wire for 6 months or until reaching a clinically acceptable little irregularity index of less than 1 mm.

7. Sample Size

Our sample size calculation is based on a study which assessed the use of nickel-titanium lingual wire for retreating relapsed lower incisors and reported a significant decrease in Little's Irregularity Index from the pretreatment values. The mean post-treatment Little's Irregularity Index was 0.8 with a standard deviation (SD) of 0.40. A minimal clinically significant difference of 0.6 was determined based on expert opinion.

Sample size calculation was conducted using Power and Sample Size (PS) software (Department of Biostatistics, Vanderbilt University). A t-test was performed with the power set to 0.8, an allocation ratio of 1:1:1, and a Type I error probability (alpha) of 0.05. The results indicated that group sample sizes of 8, 8, and 8 would achieve 90% power to detect significant differences.

To account for potential patient loss to follow-up (attrition), the sample size was increased, resulting in a total of 30 participants, with 10 participants allocated to each of the three groups.

8. Randomization

8a. Sequence generation

The randomization of the recruited subjects will be done with a randomized list, using random.org website. This list is made by an individual not involved in the clinical trial.

8b. Type

The type of randomization will be block randomization. The number of blocks and block sizes will be blinded to the investigators.

9. Allocation and concealment mechanism

Each patient will be allocated a number from sequentially numbered opaque sealed envelopes after fulfillment of the inclusion criteria and signing the informed consent to be enrolled in the study.

According to the number, the patients will be then allocated into one of the groups using a randomization table.

10. Implementation Before the beginning of the research, the allocation sequence will be generated by someone not involved in the study. The random list will be concealed from the principal investigator, who will be responsible for enrolling participants. Each participant will draw a sealed number, after which the allocation will be implemented by the person generating the sequence. All contributors to the study will remain blinded to the random list. The treatment type will be securely stored in sealed envelopes to ensure allocation concealment.

11. Blinding

Blinding will be carried out only for the data assessment because the researchers, participants and subjects can not be blinded. Therefore, a person who does not know the nature of the trial will analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate lower incisors crowding. (Little irregularity index of 3-6 mm)
* Relapse from previous non extraction orthodontic treatment that finished at least 1 year before the study.
* Patient refuses to go through full comprehensive orthodontic treatment.

Exclusion Criteria:

* Extracted or missing lower incisor or lower canine.
* Orthodontic patients who experienced relapse and were treated with extractions.
* Medically compromised patients.
* Hypersensitivity or allergy to any material involved in the study.
* Patients suffering from any congenital, hereditary or systemic disease.
* Root resorption in lower anterior teeth.
* Carious or fractured lower anterior teeth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Resolution of lower anterior teeth crowding | 6 months
  This outcome was detected through measurement of the mean change in the little irregularity index which is defined as the sum of the linear distances between the anatomical contact points of the mandibular incisors.
  The little irregularity index will be measured using 3shape ortho analyzer software.

SECONDARY OUTCOMES:
Treatment Duration | 6 months
  The treatment will be considered completed when the alignment of the lower anterior teeth reaches a clinically acceptable little irregularity index of less than 1 mm or after 6 months of treatment initiation. It will be assessed by clinical observation and recorded in weeks.
Patient expectations | 6 months
  Each patient will fill a questionnaire regarding his treatment experience in a scale from 0-5. The questionnaire will include several questions related to oral hygiene, pain and discomfort experienced throughout the trial. The questionnaire will be filled at the end of the treatment.
Pain reported on Visual analogue scale | This outcome will be recorded at 8 time points which are: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7 and Day 14.
  Each patient's level of discomfort will be assessed by a scale on which the patient marks the degree of pain on a scale from 0-10 where 0 represented no pain and 10 presented severe pain (Appendix 11). This outcome was recorded at 8 time points which are: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7 and Day 14.
Gingival inflammation | This outcome will be recorded at 4 timepoints, Pre treatment, 4 weeks after treatment, 12 weeks after treatment, Post treatment or after 6 months of treatment.
  Gingival inflammation of the lower 6 anterior teeth was assessed using Loe and Silness gingival index.The gingiva was examined at four sites around each lower anterior tooth ( From canine to canine): mesial, distal, labial, and lingual. Each site is scored based on the gingival index criteria, and the scores are averaged to provide and overall gingival index score for the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univeristy, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Franchi L, Giuntoli F, Fortini A, Chiodo BP, Baccetti T. A simplified lingual technique. J Clin Orthod. 2010 Mar;44(3):183-9. No abstract available. PMID 20575320
- [Background] Yu Y, Sun J, Lai W, Wu T, Koshy S, Shi Z. Interventions for managing relapse of the lower front teeth after orthodontic treatment. Cochrane Database Syst Rev. 2013 Sep 6;2013(9):CD008734. doi: 10.1002/14651858.CD008734.pub2. PMID 24014170
- [Background] Liou EJ, Chen LI, Huang CS. Nickel-titanium mandibular bonded lingual 3-3 retainer: for permanent retention and solving relapse of mandibular anterior crowding. Am J Orthod Dentofacial Orthop. 2001 Apr;119(4):443-9. doi: 10.1067/mod.2001.111397. PMID 11298318
- [Background] Little RM, Riedel RA, Artun J. An evaluation of changes in mandibular anterior alignment from 10 to 20 years postretention. Am J Orthod Dentofacial Orthop. 1988 May;93(5):423-8. doi: 10.1016/0889-5406(88)90102-3. PMID 3163221
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332